CLINICAL TRIAL: NCT01965782
Title: Disposition of [14C]-LY3023703 Following Oral Administration in Healthy Subjects
Brief Title: A Study of [14C]-LY3023703 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to safety results from another trial of LY3023703. No participants in this study received study drug.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15097; I6H-MC-MCBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [^14C]-LY3023703 (Experimental): Single oral dose of 15 mg LY3023703, containing approximately 100 µCi [^14C] labeled drug, administered as an oral solution.
  Interventions: Drug: [^14C]-LY3023703

INTERVENTIONS:
Drug: [^14C]-LY3023703 — Administered orally

SUMMARY:
This type of study is called a radiolabeled study. For this study, LY3023703 (study drug) has been specially prepared to contain radiolabeled carbon [14C]. [14C] is a naturally occurring radioactive form of the element carbon. This study will help understand how the drug appears in the blood, urine, and stool after it is administered to healthy men. Information about any side effects that may occur will also be collected. This study will last up to 15 days for each participant, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants will either be sterile or, if sexually active, agree to use approved methods of contraception from the day before dosing until 3 months after the follow-up assessment
* Participants will refrain from sperm donation from the day before dosing until 3 months after the follow-up assessment
* Have a body mass index (BMI) of 18.5 to 32.0 kilogram per meter square (kg/m^2)
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have given written informed consent approved by Lilly and the IRB governing the site

Exclusion Criteria:

* Are currently enrolled in, have participated, within the last 30 days, in a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Are participants who have previously completed or withdrawn from this study or any other study investigating LY3023703, and have previously received the investigational product
* Have known allergies to LY3023703, related compounds or any components of the formulation, or history of significant atopy
* Have recent or ongoing gastrointestinal (GI) symptoms or illnesses, have a history of GI bleeding or perforation, related to previous nonsteroidal anti-inflammatory drug (NSAID) or cyclooxygenase (COX)2 inhibitor therapy or have active or history of recurrent peptic ulcer/hemorrhage (2 or more distinct episodes of proven ulceration or bleeding)
* Have a history of intolerance to NSAIDs or aspirin
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of alanine aminotransferase or aspartate aminotransferase levels above the normal ranges, confirmed on repeat, or a history of elevated and abnormal liver tests
* Have intended use of over-the-counter medications or prescription medication within 14 days prior to dosing. Also within 30 days prior to dosing, any drugs and dietary items that are known inducers or inhibitors of cytochrome P450 (CYP) 3A or CYP2J2 or other drugs that may affect the disposition of LY3023703 or increase risk for complications from the study
* Have consumed herbal supplements within 14 days prior to admission or grapefruit juice, grapefruits, grapefruit-containing products, Seville orange juice, Seville oranges, star fruit, or star fruit juice within 7 days prior to dosing or intend to consume during the study
* Have donated blood of more than 500 milliliter (mL) within the last month
* Have participated in a [14C]-study within the last 6 months prior to admission for this study
* Exposure to significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)
* A positive alcohol breathalyzer test
* A positive cotinine test
* Are unwilling to refrain from consuming xanthine-containing food and drink from 48 hours prior to admission until discharge from the Clinical Research Unit (CRU)
* Have a defecation pattern less than once per 2 days or acute constipation within 3 weeks of the day before dosing
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 subjects were screened and enrolled but no drug was given or other data collected due to the study being terminated.
Groups:
- [^14C]-LY3023703: Single dose of 15 mg LY3023703, containing approximately 100 µCi [^14C] labeled drug, administered as an oral solution.
Period: Overall Study
Arm/Group | [^14C]-LY3023703
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 18 subjects were screened and enrolled but no drug was given or other data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Fecal Excretion of LY3023703 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Time Frame: Predose up to 168 hours post dose
Population: No drug was given or data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Number analyzed (Participants) | 0

2. Primary Outcome: Urinary Excretion of LY3023703 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Time Frame: Predose up to 168 hours post dose
Population: No drug was given or data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Number analyzed (Participants) | 0

3. Secondary Outcome: Pharmacokinetics of LY3023703 and Radioactivity Maximum Observed Concentration (Cmax)
Time Frame: Predose up to 168 hours post dose
Population: No drug was given or data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Number analyzed (Participants) | 0

4. Secondary Outcome: Pharmacokinetics of LY3023703 and Radioactivity Time of Maximum Observed Concentration (Tmax)
Time Frame: Predose up to 168 hours post dose
Population: No drug was given or data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Number analyzed (Participants) | 0

5. Secondary Outcome: Pharmacokinetics of LY3023703 and Radioactivity Area Under The Concentration-Time Curve From Time Zero to the Last Timepoint With a Measurable Concentration [AUC (0 to Tlast)]
Time Frame: Predose up to 168 hours post dose
Population: No drug was given or data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Number analyzed (Participants) | 0

6. Secondary Outcome: Relative Abundance of LY3023703 and the Metabolites of LY3023703 in Urine and Feces
Time Frame: Predose up to 168 hours post dose
Population: No drug was given or data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Number analyzed (Participants) | 0

7. Secondary Outcome: Relative Abundance of LY3023703 and the Metabolites of LY3023703 in Plasma
Time Frame: One hour post-dose up to 72 hours post dose
Population: No drug was given or data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No drug was given or data collected due to the study being terminated.
Arm/Group | [^14C]-LY3023703
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
18 subjects were screened and enrolled but no drug was given or other data collected due to the study being terminated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days